CLINICAL TRIAL: NCT00290602
Title: Prospective Phase II Study of Early Low Dose Steroid Therapy of Acute Respiratory Distress Syndrome (ARDS) After Thoracic Surgery (E-START)
Brief Title: Early Low Dose Steroid Therapy of Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-04-087
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury; Postoperative Complications
Keywords: Acute respiratory distress syndrome; corticosteroids; postoperative complications; cytokines
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Postoperative Complications | interventions — Methylprednisolone Hemisuccinate

INTERVENTIONS:
Drug: Methylprednisolone sodium succinate

SUMMARY:
The purpose of this study is to determine whether the 2mg/kg administration of corticosteroids, in the form of methylprednisolone sodium succinate, in early phase acute respiratory distress syndrome after thoracic surgery, will reduce the postoperative mortality.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) developing after thoracic surgery is usually a lethal complication. The use of corticosteroid in ARDS has been the subject of great controversy and debate over the years. Unfortunately, trials of short-term, high-dose steroid therapy failed to show an improvement in mortality of patients at risk of, or with early, ARDS. Several investigators have suggested that the use of corticosteroids in the late or fibroproliferative phase of ARDS improved lung function and survival.

Recently some authors have demonstrated that there is a potential for pulmonary fibroproliferation during the early stages of ARDS and the use of low-dose corticosteroids at these early stages has been found to lead to a complete maintenance of in vivo and in vitro respiratory mechanics in acute lung injury. These articles had important implications both for the study of repair mechanisms and the timing of therapies.

ELIGIBILITY:
Inclusion Criteria:

1. ARDS, defined as the acute onset of:

   * PaO2/FiO2 ≤ 200.
   * Bilateral infiltrates. The infiltrates may be patchy, diffuse, homogeneous, or asymmetric, and should be consistent with pulmonary edema or the fibrotic changes of fibroproliferation. Opacities due to pleural effusions or atelectasis should not be considered. If pneumonectomy, unilateral infiltrate is included.
   * No evidence of left atrial hypertension. If measured, PAWP ≤ 18 mmHg.
   * Criteria a-c must occur together within a 24-hour interval. The first date that these criteria are met is defined as the onset of ARDS
2. Since ARDS onset, chest infiltrates must be progressive, and chest computed tomographic scan findings are consistent with postoperative ARDS findings or ground glass opacities by radiologists.
3. Major thoracic surgery

   * Lung cancer; pneumonectomy, extended pneumonectomy, lobectomy, sleeve lobectomy, extended lobectomy, wedge resection.
   * Esophageal cancer; Ivor-Lewis operation, transhiatal esophagectomy, McKeown operation.
   * Metastatic lung cancer; simultaneous bilateral metastasectomy.
4. PaO2/FiO2 ≤ 200 on the day of E-START enrollment.

Exclusion Criteria:

1. Clinical evidence of active and untreated infection.

   Clarifications:
   * A known, undrained abscess (e.g. Staphylococcal lung abscess or loculated empyema or intra-abdominal abscess) or a known intravascular nidus of infection (e.g., bacterial or fungal endocarditis) will be a basis for exclusion, even if it is being treated with antibiotics.
   * A bacterial infection being treated with a standard antibiotic regimen would not be a basis for exclusion.
   * Disseminated fungal infection, even if being treated, is an exclusion.
   * Ongoing septic shock, even if on antibiotics is a basis for exclusion.
2. Age <18 years.
3. Pregnancy.
4. Burns requiring skin grafting.
5. Patients with AIDS by CDC criteria, diagnosed by either a documented AIDS defining illness or CD4<200(see Appendix F); prednisolone therapy >=300mg(or its equivalent) cumulative dose within 21 days prior to enrollment, or >15mg/day(or its equivalent) within 7 days prior to enrollment; cytotoxic therapy within 3 weeks.
6. Other irreversible chronic disease or condition for which 6 month mortality is estimated ≥ 50%.
7. Not committed to full support.
8. Severe chronic liver disease (Child-Pugh Class C score>10 points).
9. Transplant patients with the exception of autologous bone marrow transplants.
10. Extracorporeal support of gas exchange at the time of study entry (e.g., ECMO).
11. Known or suspected adrenal insufficiency.
12. Vasculitis with diffuse alveolar hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-02; Study Completion 2006-12

PRIMARY OUTCOMES:
the percentage of patients alive at postoperative 30 day; Patients discharged alive from the hospital in unassisted breathing before 60 days

SECONDARY OUTCOMES:
the percentage of ventilator-free patients at 7 days from study entry; the percentage of oxygen-independent patients at 21 days following study entry; response of inflammatory mediators to the novel treatment; pulmonary function in ARDS survivors

CONTACTS AND LOCATIONS:
Overall Officials: Jae Ill Zo, MD, PhD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Lee HS, Lee JM, Kim MS, Kim HY, Hwangbo B, Zo JI. Low-dose steroid therapy at an early phase of postoperative acute respiratory distress syndrome. Ann Thorac Surg. 2005 Feb;79(2):405-10. doi: 10.1016/j.athoracsur.2004.07.079. PMID 15680804
- [Background] Annane D, Sebille V, Bellissant E; Ger-Inf-05 Study Group. Effect of low doses of corticosteroids in septic shock patients with or without early acute respiratory distress syndrome. Crit Care Med. 2006 Jan;34(1):22-30. doi: 10.1097/01.ccm.0000194723.78632.62. PMID 16374152
- See also: ARDS network — http://www.ardsnet.org
- See also: National Cancer Center Korea — http://www.ncc.re.kr